CLINICAL TRIAL: NCT02295943
Title: Objective Evaluation of Postoperative Positioning in Macular Hole Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not meet primary and secondary outcome measures
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Haukeland University Hospital (Other); Trondheim University Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/879
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Macular Hole
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positioning measuring device (Other): The supine time during the first postoperative day is measured
  Interventions: Other: Positioning measuring device

INTERVENTIONS:
Other: Positioning measuring device — Vitrectomy, intraocular gas fill. The supine time during the first postoperative day is measured

SUMMARY:
The macular hole formation takes place in the centre of the retina. A closure of the macular hole is believed to take place if the central retinal area is kept dry in the postoperative period. Therefore the eye is filled with a gas mix and the patients are urged to avoid the supine position in the first postoperative days. The investigators have developed a positioning measuring device which can measure the extent of supine positioning time. Patients are to carry the positioning measuring device during the first postoperative 24 hours. Hereby the investigators search new knowledge concerning patients compliance and its relation to macular hole closure.

ELIGIBILITY:
Inclusion Criteria:

* Primary macular hole
* Duration less than 24 months
* Informed consent

Exclusion Criteria:

* Secondary macular hole i.e. trauma, excessive myopia (more than 6 dioptres)
* Previous vitreomacular surgery
* Age under 18 years
* Unable to sign

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Macular hole closure | 2 weeks

SECONDARY OUTCOMES:
Time in supine sleeping position | 1 day after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Forsaa, MD, Principal Investigator — Stavanger University Hospital, Department of Ophthalmology
Locations (4):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindtjorn B, Krohn J, Austeng D, Fossen K, Varhaug P, Basit S, Helgesen OH, Eide GE, Forsaa VA. Nonsupine Positioning after Macular Hole Surgery: A Prospective Multicenter Study. Ophthalmol Retina. 2019 May;3(5):388-392. doi: 10.1016/j.oret.2018.12.006. Epub 2018 Dec 31. PMID 31044728